CLINICAL TRIAL: NCT02855775
Title: Study of the Relative Impact of the Neonatal Fc Receptor (FcRn) and the Therapeutic History on Monoclonal Antibodies Elimination. Proof of the Concept on Patients Treated by Bevacizumab or Trastuzumab in Breast Cancer
Brief Title: Monoclonal Antibodies Elimination in Breast Cancer Patient
Acronym: PK-MAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: API/2011/21
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab (Experimental): Bevacizumab in monotherapy or in association to other anticancer agents pharmacokinetic assessment with blood sample with additional blood sample
  Interventions: Other: additional blood sample
- Trastuzumab (Experimental): Trastuzumab in monotherapy or in association to other anticancer agents pharmacokinetic assessment with blood sample with additional blood sample
  Interventions: Other: additional blood sample

INTERVENTIONS:
Other: additional blood sample — blood sample every 3 weeks

SUMMARY:
This Study evaluates covariables being able to potentially influence the elimination of the monoclonal antibodies (trastuzumab, bevacizumab and denosumab).

DETAILED DESCRIPTION:
Monoclonal antibodies are very widely used in cancer treatment . Certain patients benefit from these antibodies for several years and it is conceivable to wonder about the evolution of the pharmacokinetics of these antibodies.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosed cancer
* patient treated by bevacizumab or trastuzumab
* Life expectancy of at least 3 months
* For the women: menopausal women for at least 24 months, sterilized surgically, or, for the women old enough to procreate, use a method of effective contraception (oral contraceptives, contraceptive injections, intra-uterine devices, method of the double barrier, the contraceptive patches). This contraception will have to be pursued during 6 months after the end of the treatment by bevacizumab or by trastuzumab.

Exclusion Criteria:

* For Patients treated by trastuzumab: Dyspnoea of severe rest in touch with complications due to the disease or requiring an oxygen therapy.
* Hypocalcemia severe untreated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
clearance of the bevacizumab | 9 months

SECONDARY OUTCOMES:
clearance of the trastuzumab | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No